CLINICAL TRIAL: NCT00987636
Title: Phase 3, Open Label, Multi-centre, Randomised Controlled International Study in Ewing Sarcoma
Brief Title: Study in Localized and Disseminated Ewing Sarcoma
Acronym: EWING2008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108128; 2008-003658-13 (EudraCT Number)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Ewing's Sarcoma
Keywords: Ewing Sarcoma; localized; disseminated; metastases; bone; soft tissue
MeSH Terms: conditions — Sarcoma, Ewing; Neoplasm Metastasis | interventions — Zoledronic Acid; Diphosphonates; Busulfan; treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- R1 (Experimental): Standard Risk R1: in a randomised trial, to examine whether add-on treatment with zoledronic acid in addition to induction and maintenance chemotherapy improves event-free survival in patients with localised Ewing sarcoma and good histological response or with initial tumour volume <200 mL compared to no add-on treatment.
  Interventions: Drug: Zoledronic acid
- R2 (Experimental): High Risk R2: in a randomised trial, to examine whether high-dose chemotherapy using busulfan-melphalan with autologous stem cell reinfusion, compared with standard chemotherapy, improves event-free survival in patients with localised Ewing sarcoma and poor histological response or tumour volume ≥200 mL (R2loc). In patients with pulmonary metastases high dose busulfan-melphalan chemotherapy with autologous stem cell reinfusion is randomised versus standard chemotherapy plus whole lung irradiation (R2pulm).
  Interventions: Drug: Busulfan
- R3 (Experimental): Very High Risk R3: in a randomised trial, to examine whether the addition of high dose chemotherapy using treosulfan-melphalan followed by autologous stem cell reinfusion to eight cycles of standard adjuvant chemotherapy, compared to eight cycles of standard adjuvant chemotherapy alone, improves event-free survival in patients with primary disseminated disease.
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Zoledronic acid — intravenously at 28 day intervals beginning with cycle 6 of VAC/VAI consolidation chemotherapy for a total period of nine months.
  Patients < 18 years will receive 0.05 mg/kg BW by IV infusion 30 min-1 h.
  Patients >= 18 years will receive a bodyweight-dependent dose:
  Patients >40kg receive 4 mg by IV infusion 30 min-1h Patients 20-40 kg receive 2 mg by IV infusion 30 min-1h
  Other Names: Zometa; Bisphosphonate
  Arms: R1
Drug: Busulfan — intravenously, day -6 to d -3 adults: 0.8 mg/kg body weight (BW) children and adolescents: <9 kg= 1mg/kg BW 9 - <16 kg= 1.2 mg/kg BW 16 - 23 kg= 1.1 mg/kg BW >23 - 34 kg= 0.95 mg/kg BW >34 kg = 0.8 mg/kg BW
  Other Names: Busilvex
  Arms: R2
Drug: Treosulfan — 12 g/m² d-5 to d-3
  Arms: R3

SUMMARY:
Ewing Sarcoma

Primary objectives:

Standard Risk R1: in a randomised trial, to examine whether add-on treatment with zoledronic acid in addition to induction and maintenance chemotherapy improves event-free survival in patients with localised Ewing sarcoma and good histological response or with initial tumour volume <200 mL compared to no add-on treatment.

*High Risk R2: in a randomised trial, to examine whether high-dose chemotherapy using busulfan-melphalan with autologous stem cell reinfusion, compared with standard chemotherapy, improves event-free survival in patients with localised Ewing sarcoma and poor histological response or tumour volume ≥200 mL (R2loc). In patients with pulmonary metastases high dose busulfan-melphalan chemotherapy with autologous stem cell reinfusion is randomised versus standard chemotherapy plus whole lung irradiation (R2pulm).

Very High Risk R3: in a randomised trial, to examine whether the addition of high dose chemotherapy using treosulfan-melphalan followed by autologous stem cell reinfusion to eight cycles of standard adjuvant chemotherapy, compared to eight cycles of standard adjuvant chemotherapy alone, improves event-free survival in patients with primary disseminated disease.

*R2 accrual discontinued on December 1st 2015.

DETAILED DESCRIPTION:
EWING 2008 is a joint protocol of European and North American Ewing sarcoma study groups. The protocol is aimed at optimising treatment and treatment results of patients with Ewing sarcomas. The EWING 2008 protocol is open to all patients diagnosed with Ewing sarcomas, localised or metastatic, who are considered eligible for neoadjuvant chemotherapy. All patients registered will receive induction chemotherapy consisting of six cycles of vincristine, ifosfamide, doxorubicin and etoposide (VIDE). The decision regarding local therapy must be made following the fifth cycle of induction treatment, with a preference for surgical intervention with or without additional radiotherapy. Preoperative radiotherapy may be considered to improve the operability of otherwise inoperable lesions. In patients with localised disease or with pulmonary metastases, local treatment should be performed following the 6th cycle of VIDE chemotherapy, and should be a complete tumour resection, whenever feasible. Post-operative radiotherapy is determined by the completeness of surgery and the histological response to chemotherapy.

Standard Risk R1 Good responders (R1) (< 10% viable tumour cells) with localised disease are allocated to the standard risk arm and will receive a further eight cycles of chemotherapy composed of vincristine, actinomycin D, and cyclophosphamide (VAC) (females) or ifosfamide instead of cyclophosphamide (VAI) (males). They will be randomised to receive add-on treatment with either fenretinide, zoledronic acid, fenretinide plus zoledronic acid, or no add-on treatment.

High Risk R2 *Poor responders (R2) with localised disease will continue to be randomised as in EURO-E.W.I.N.G. 99 to receive either eight cycles of VAI chemotherapy or high dose treatment with busulfan-melphalan (R2loc).

Patients with primary pulmonary metastases are also allocated to continue to be randomised as in EURO-E.W.I.N.G. 99 to receive either eight cycles of VAI chemotherapy or high dose treatment with busulfan-melphalan (R2pulm).

Very High Risk R3 Patients with disseminated disease, i.e. dissemination to bone and/or other sites and possibly additional pulmonary dissemination (R3), receive six cycles of VIDE induction chemotherapy. Patients are then randomised to either continue with eight cycles of vincristine, actinomycin D and cyclophosphamide (VAC) chemotherapy or high dose treosulfan-melphalan (TreoMel) chemotherapy followed by autologous stem cell reinfusion followed thereafter by eight cycles of VAC chemotherapy. Local therapy in R3 patients is following VIDE induction, whenever feasible prior to high dose therapy (HDT). When long periods of immobilisation following surgery are anticipated, e.g pelvic reconstruction, surgery following HDT may be advisable. Depending on clinical response to induction chemotherapy radiotherapy prior to HDT and surgery may be an option to be considered in such patients. Any delay between VIDE and HDT for reasons of e.g. local treatment must be bridged with VAC cycles. The total number of VAC cycles is not to exceed eight cycles.

*R2 accrual discontinued on December 1st 2015.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed Ewing sarcoma of bone or soft tissue.
* Age and sex: Either sex, age >48 months (for GPOH patients) and <50 years at the date of diagnostic biopsy. Younger or elderly patients may be reported to the appropriate office (see section 1.4) but are not included in this study.
* Registration: ≤ 45 days after diagnostic biopsy/surgery.
* Start of chemotherapy: ≤ 45 days after diagnostic biopsy/surgery.
* Informed consent: Must be signed prior to study entry.
* Performance status: Lansky or Karnofsky score > 50%, may be modified for handicapped patients.
* Haematological parameters:

  * Haemoglobin > 8 g/dl (transfusion allowed),
  * Platelets > 80.000/µl (transfusion allowed),
  * WBC > 2000/µl.
* Cardiac values: LVEF > 40%, SF > 28%.

Exclusion Criteria:

* More than one cycle of other chemotherapy prior to registration
* Second malignancy
* Pregnancy and lactation
* Concurrent treatment within any other clinical trial, except trials with different endpoints that due to the nature of their endpoints must run parallel to EWING 2008 e.g. trials on antiemetics, antimycotics, antibiotics, strategies for psychosocial support, etc...
* Any other medical, psychiatric, or social condition incompatible with protocol treatment

Ages: 48 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 907 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Event free survival | 9.5 years

SECONDARY OUTCOMES:
Overall survival | 9.5 years
Safety and toxicity | permanent
Quality of life | 9.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Uta Dirksen, Prof MD, Principal Investigator — University Hospital, Essen; Alan W Craft, Prof Sir MD, Study Chair — Royal Victoria Infirmary; Heribert Jürgens, Prof MD, Study Chair — University Hospital Muenster
Locations (2):
- Germany (2):
  - University Hopital Essen, Pediatrics III, Hematology/ Oncology, Sarcoma Centre, International Ewing Sarcoma Study Group, West German Cancer Centre, Essen
  - University Children´s Hospital, Pediatric Hematology and Oncology, Münster

REFERENCES:
- [Derived] Stork T, Ranft A, Aigner C, Jurgens H, Ladenstein RL, Timmermann B, Van den Berg H, Dirksen U, Collaud S. Primary Mediastinal Ewing's Sarcoma: Post Hoc Analysis from Two International Multicenter Prospective Randomized Trials. Cancers (Basel). 2025 Jan 2;17(1):118. doi: 10.3390/cancers17010118. PMID 39796745
- [Derived] Rechl V, Ranft A, Bhadri V, Brichard B, Collaud S, Cyprova S, Eich H, Ek T, Gelderblom H, Hardes J, Haveman LM, Hartmann W, Hauser P, Heesen P, Jurgens H, Kanerva J, Kuhne T, Raciborska A, Rascon J, Streitburger A, Uhlenbruch Y, Timmermann B, Kersting J, Pham MT, Dirksen U. Factors Influencing the Outcome of Patients with Primary Ewing Sarcoma of the Sacrum. Sarcoma. 2024 Mar 16;2024:4751914. doi: 10.1155/2024/4751914. eCollection 2024. PMID 38524902
- [Derived] Koch R, Gelderblom H, Haveman L, Brichard B, Jurgens H, Cyprova S, van den Berg H, Hassenpflug W, Raciborska A, Ek T, Baumhoer D, Egerer G, Eich HT, Renard M, Hauser P, Burdach S, Bovee J, Bonar F, Reichardt P, Kruseova J, Hardes J, Kuhne T, Kessler T, Collaud S, Bernkopf M, Butterfass-Bahloul T, Dhooge C, Bauer S, Kiss J, Paulussen M, Hong A, Ranft A, Timmermann B, Rascon J, Vieth V, Kanerva J, Faldum A, Metzler M, Hartmann W, Hjorth L, Bhadri V, Dirksen U. High-Dose Treosulfan and Melphalan as Consolidation Therapy Versus Standard Therapy for High-Risk (Metastatic) Ewing Sarcoma. J Clin Oncol. 2022 Jul 20;40(21):2307-2320. doi: 10.1200/JCO.21.01942. Epub 2022 Apr 15. PMID 35427190
- [Derived] Dirksen U, Brennan B, Le Deley MC, Cozic N, van den Berg H, Bhadri V, Brichard B, Claude L, Craft A, Amler S, Gaspar N, Gelderblom H, Goldsby R, Gorlick R, Grier HE, Guinbretiere JM, Hauser P, Hjorth L, Janeway K, Juergens H, Judson I, Krailo M, Kruseova J, Kuehne T, Ladenstein R, Lervat C, Lessnick SL, Lewis I, Linassier C, Marec-Berard P, Marina N, Morland B, Pacquement H, Paulussen M, Randall RL, Ranft A, Le Teuff G, Wheatley K, Whelan J, Womer R, Oberlin O, Hawkins DS; Euro-E.W.I.N.G. 99 and Ewing 2008 Investigators. High-Dose Chemotherapy Compared With Standard Chemotherapy and Lung Radiation in Ewing Sarcoma With Pulmonary Metastases: Results of the European Ewing Tumour Working Initiative of National Groups, 99 Trial and EWING 2008. J Clin Oncol. 2019 Dec 1;37(34):3192-3202. doi: 10.1200/JCO.19.00915. Epub 2019 Sep 25. PMID 31553693
- [Derived] van den Berg H, Paulussen M, Le Teuff G, Judson I, Gelderblom H, Dirksen U, Brennan B, Whelan J, Ladenstein RL, Marec-Berard P, Kruseova J, Hjorth L, Kuhne T, Brichard B, Wheatley K, Craft A, Juergens H, Gaspar N, Le Deley MC; Euro-EWING99 Group. Impact of gender on efficacy and acute toxicity of alkylating agent -based chemotherapy in Ewing sarcoma: secondary analysis of the Euro-Ewing99-R1 trial. Eur J Cancer. 2015 Nov;51(16):2453-64. doi: 10.1016/j.ejca.2015.06.123. Epub 2015 Aug 10. PMID 26271204